CLINICAL TRIAL: NCT01216722
Title: Comparison of Targeted Lower Extremity Strengthening and Usual Care Progressive Ambulation in Subjects Post Liver Transplant: A Randomized Controlled Trial
Brief Title: Study of Resistance Strengthening Versus Ambulation Post-Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: David Mandel, Investigator, University of Miami Dept. of Physical Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070787
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-07

CONDITIONS: Liver Transplantation; Resistance Training; Activities of Daily Living
Keywords: Muscle Wasting; Strengthening; Liver Disease; Transplant
MeSH Terms: conditions — Muscular Atrophy; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Strengthening (Experimental): Body weight antigravity positioning and elastic resistance bands are used to provide resistance for strengthening in supine, sitting, and standing in subjects post liver transplant.
  Interventions: Other: Resistance Strengthening Exercise Program
- Usual Care Control (No Intervention): Subjects perform the usual care of progressive ambulation and increased activity post liver transplant

INTERVENTIONS:
Other: Resistance Strengthening Exercise Program — Home exercise Program. 3-4 days a week. 30 minutes a session. 12 weeks
  Arms: Resistance Strengthening

SUMMARY:
Resistance strengthening exercise will increase strength and functional activity greater than ambulation in subjects post-liver transplantation.

DETAILED DESCRIPTION:
Individuals post liver transplantation are significantly muscle wasted due to chronic liver disease. Current Usual care only involves progressive ambulation. Resistance exercise targeted at the lower extremities are anticipated to increase muscle strength in the muscles that extend the hip, extend the knee, and plantar flex the ankle more than seen with the usual care ambulation. The anticipated increases in strength should improve functional performance of activities such as standing from a chair, walking, and climbing stairs. The improvement in strength and functional performance should improve an individuals quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Undergone Liver Transplantation a minimum of 6 weeks and a maximum of 12 weeks prior to enrollment
* Ambulatory without physical assistance, but permitted to use a cane or walker

Exclusion Criteria:

* Diagnosis of Hepatocellular Carcinoma
* Significant Cardiopulmonary disease
* Neurological / Neuromuscular Disorder including cerebral vascular accident (CVA), Parkinson's Disease, Alzheimer's Disease, Dementia unrelated to Hepatic Encephalopathy, dystonia, multiple sclerosis, and polio.
* Blindness
* Inability to comprehend the English or Spanish Language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Baseline
Heel Rise Test | Baseline
30-Second Chair-Stand Test | Baseline
Bridge Test | Baseline
Six Minute Walk Test | 12 weeks
Heel Rise Test | 12 weeks
30-Second Chair-Stand Test | 12 weeks
Bridge Test | 12 weeks

SECONDARY OUTCOMES:
Short Form (SF-36) Questionnaire | Baseline
Short Form (SF-36) Questionnaire | 12 weeks
Chronic Liver Disease Questionnaire (CLDQ) | Baseline
Chronic Liver Disease Questionnaire (CLDQ) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Roach, PhD, PT, Study Chair — University of Miami; David W Mandel, PhD, PT, Principal Investigator — University of Miami Dept. of Physical Therapy
Locations (1):
- University of Miami Department of Physical Therapy, Coral Gables, Florida, United States